CLINICAL TRIAL: NCT04541862
Title: Adult Intensive Care Units Database of National Taiwan University Hospital
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201901010RIND
Record Dates: First submitted 2020-08-30; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients
  Interventions: Other: Intensive care

INTERVENTIONS:
Other: Intensive care — intensive care for critically ill patients in the intensive care units

SUMMARY:
Australian and New Zealand Intensive Care Society (ANZICS) has built an Center of Outcome and Resource Evaluation (CORE) adult patients database (APD) of adult critically ill patients. ANZICS CORE APD has built an international collaboration of intensive care unit (ICU) database. National Taiwan University Hospital has joined this international collaboration and built the data according to the APD data dictionary with same value domain attributes and data element attributes. This database also add expansion of data include hourly vital signs data, more laboratory data, more diagnoses at admission and discharge, data after 24 hours till discharge, and extended information of clinical outcomes more than 30 days after admission to ICU .

This database will retrospectively collect the data of patients discharged from intensive care after March 1, 2019 and will prospectively continue the retrospective collection of data till the patients discharged before June 30, 2043.

The data will be used for the evaluation of quality and resource allocation, quality improvement, education of data science, datathon, and research to predict the clinical outcomes and assist the treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients admitted to intensive care units

Exclusion Criteria:

* Patients aged less than 20 years

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to intensive care units.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2043-06 (Estimated); Study Completion 2043-12 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  Survival status at 30 days after ICU admission

SECONDARY OUTCOMES:
Length of stay in intensive care unit | Time to discharge from intensive care unit, a median of 2-7 days
  Length of stay (days) in intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available according to the regulation of Research Ethic Committee of National Taiwan University Hospital.